CLINICAL TRIAL: NCT01330940
Title: Effect of Diet Orange Soda on Urinary Lithogenicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, David S. Goldfarb, M.D., Chief, Nephrology, VA New York Harbor Healthcare System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1100
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Stones; Nephrolithiasis; Urolithiasis
Keywords: Kidney stones; Calcium; citrate
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water drinking (Placebo Comparator): 32 ounces of water/24 hours
  Interventions: Dietary Supplement: Orange soda
- orange soda drinking (Active Comparator): 32 ounces orange soda
  Interventions: Dietary Supplement: Orange soda

INTERVENTIONS:
Dietary Supplement: Orange soda — 32 ounces per day

SUMMARY:
Beverages containing citrate may be useful in increasing urine citrate content and urine pH. Such changes in urine chemistry could help prevent kidney stones. Diet orange soda has more citrate than other similar beverages. The investigators are interested in whether diet soda will improve urine chemistry in the appropriate manner.

DETAILED DESCRIPTION:
The effect of orange soda compared with water in changing 24 hour urine citrate excretion in mg/day will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* able to sign consent
* ability to reliably urinate into a vessel and measure urine volume

Exclusion Criteria:

* prior history of nephrolithiasis
* a known history of metabolic bone disease
* hyperthyroidism
* hyperparathyroidism or chronic kidney disease
* current use of diuretics
* current use of potassium citrate or other oral alkali supplementation and
* use of calcium supplementation that could not be stopped

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in urine citrate content | 1 week
  Citrate is measured in 24h urine sample and expressed as mg/day

SECONDARY OUTCOMES:
Change in urine pH | One week
  urine pH is measured in a 24h urine sample and has no units

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Principal Investigator — New York Harbor VA Medical Center
Locations (1):
- New York Harbor VA Medical Center, New York, New York, United States